CLINICAL TRIAL: NCT03591497
Title: Role of Virtual Reality in Improving Balance in Patients With Myelopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dhritiman Chakrabarti, Assistant Professor, National Institute of Mental Health and Neuro Sciences, India
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC (BS & NS DIV)/2017-18
Record Dates: First submitted 2018-06-20; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Myelopathy; Virtual Reality
Keywords: Myelopathy; Virtual Reality; Rehabilitation; Balance
MeSH Terms: conditions — Spinal Cord Diseases

STUDY DESIGN:
Intervention Model Description: Prospective Cohort study involving cases with use of intervention. Matched control cohort subjects were selected using pre-specified matching criteria (for matching with interventional cohort) as comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Instrument to be used:
  Software Neuro@home (semi immersive virtual reality system for neurological rehabilitation) was used. In each of the sessions, an avatar on screen that representing the patient was regulated by the patient to perform a virtual task that focused on the training of a specific body part.
  Programme schedule:
  Each session of virtual reality therapy lasted for thirty minutes. Day 0 included an orientation to the machine with five minutes of gaming. This was followed by virtual reality therapy for five days a week at the same time of the day for three consecutive weeks.
  Interventions: Other: Virtual Reality
- Control Group (No Intervention): Virtual reality sessions were not provided.

INTERVENTIONS:
Other: Virtual Reality — As described in Experimental arm description.
  Arms: Intervention Group

SUMMARY:
Balance of the body is achieved by the coordination of three major systems, visual, vestibular and proprioceptive sensation and by the reflexive control of the limbs. In myelopathy, factors like balance and posture, range of motion, muscle strength, coordinated motor control, muscle tone and proprioception are affected. Balance and gait rehabilitation is an important goal in myelopathy. Virtual reality (VR) is a computer based technology that is used for task oriented biofeedback therapy in rehabilitation. This study was envisioned to observe the utility of VR in rehabilitation for improving balance in patients of myelopathy.

DETAILED DESCRIPTION:
Balance of the body is achieved by the coordination of three major systems, visual, vestibular and proprioceptive sensation and by the reflexive control of the limbs. Static balance which determines the ability to maintain postural stability during sitting or standing is important to perform daily functional activities. Dynamic balance on the other hand is the ability to respond and adjust to a moving floor or any external stimuli or perturbation and is a requirement for successful gait performance.

In myelopathy, factors like balance and posture, range of motion, muscle strength, coordinated motor control, muscle tone and proprioception are affected. Lack of normal postural synergy and sensory motor integration of lower limbs and trunks and spatial information that regulate upright position and sitting balance leads to balance dysfunction in the population. Hence patient develops compensatory strategies. But ambulation involves the intricate coordination of leg movements, regulating upright posture and balance and adaptation to environmental changes. Hence balance and gait rehabilitation is an important goal in myelopathy.

Virtual reality (VR) is a computer based technology that is used for task oriented biofeedback therapy in rehabilitation. It constructs a virtual environment resembling a situation in the real world and provides multimodal sensory cues. VR ranges from non immersive to semi immersive to fully immersive, depending on the degree to which the user is isolated from the physical surroundings when interacting with the virtual environment.

In virtual reality training, participants perform functional stretching of their extremities, learn postural control of the trunk and practice weight shifting. As the level of difficulty and speed are increased for various tasks, the movement of the body's center of gravity beyond the base of support increases thus increasing the proprioceptive sensations to the joints and improves the subject's ability to adjust balance. Hence it encourages dynamic motions and functional mobility. The VR environment can be controlled and manipulated in advance to fine tune the exercises and meet individual needs. It is interactive as well as enjoyable.

Studies indicate that spinal reflex circuitry exhibits activity dependent plasticity (the capacity of the nervous system to modify its organization). Intensive task specific training is one of the most effective ways to promote neuroplasticity and develop more normalized movement patterns. VR uses this principle of neuroplasticity to promote motor relearning. Literature supports the use of VR as an effective rehabilitative tool in individuals with stroke, spinal cord injury, cerebral palsy, multiple sclerosis and other neurological disorders.

There are few studies on balance rehabilitation in myelopathy from this part of the world. Due to absence of any guidelines, identifying the most suitable type of VR system, defining the most appropriate treatment dosing, timing and intensity of training for the therapeutic application is a challenge. This study was envisioned to observe the utility of VR in rehabilitation for improving balance in patients of myelopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with myelopathy with neurological level of injury below C4.
2. Both traumatic and non-traumatic myelopathy.
3. Duration of illness less than 6 months.

Exclusion Criteria:

1. Severe orthopedic or medical impairment that interfered with sitting.
2. Upper limb muscle power <3/5.
3. Cognitive or visual impairment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Berg Balance Scale (BBS) | At admission and at discharge from hospital or 24 weeks, whichever is earlier.
  Scale is used to measure balance during functional activities. It is a 14 item scale. A 5 point scale is used for each item (0-4). "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 56. Total score is obtained by adding the individual scores.
Change in Tinetti performance oriented mobility assessment (POMA) | At admission and at discharge from hospital or 24 weeks, whichever is earlier.
  Balance section of Tinetti Performance Oriented Mobility Assessment (Tinetti Performance Oriented Mobility Assessment has two subscales, Balance and Gait section.) Balance section has 9 items. Each item can be scored in a 3 point ordinal scale (0-2). "0" indicates the lowest level of function and "2" the highest level of function. Total Score = 16. Total score is obtained by adding the individual scores.
Change in Functional reach test (forward and lateral) | At admission and at discharge from hospital or 24 weeks, whichever is earlier.
  Functional reach score. It is used to measure postural stability and dynamic balance in sitting position. It has three subsections. Right lateral reach, left lateral reach and forward lateral reach. The value of each is obtained by measuring the distance in centimeter. The total score is obtained by adding the scores of the three subsections. Lower value indicates the lower level of function and higher value the higher level of function.

SECONDARY OUTCOMES:
Difference in Berg Balance Scale (BBS) between groups | At admission and at discharge from hospital or 24 weeks, whichever is earlier.
  Scale is used to measure balance during functional activities. It is a 14 item scale. A 5 point scale is used for each item (0-4). "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 56. Total score is obtained by adding the individual scores.
Difference in Tinetti performance oriented mobility assessment (POMA) between groups | At admission and at discharge from hospital or 24 weeks, whichever is earlier.
  Balance section of Tinetti Performance Oriented Mobility Assessment (Tinetti Performance Oriented Mobility Assessment has two subscales, Balance and Gait section.) Balance section has 9 items. Each item can be scored in a 3 point ordinal scale (0-2). "0" indicates the lowest level of function and "2" the highest level of function. Total Score = 16. Total score is obtained by adding the individual scores.
Difference in Functional reach test (forward and lateral) between groups | At admission and at discharge from hospital or 24 weeks, whichever is earlier.
  Functional reach score. It is used to measure postural stability and dynamic balance in sitting position. It has three subsections. Right lateral reach, left lateral reach and forward lateral reach. The value of each is obtained by measuring the distance in centimeter. The total score is obtained by adding the scores of the three subsections. Lower value indicates the lower level of function and higher value the higher level of function.
Difference in Hospital anxiety and depression scale (HADS) between groups | At admission and at discharge from hospital or 24 weeks, whichever is earlier.
  Hospital anxiety and depression scale. It is a self-assessment scale used to detect anxiety and depression of patients under investigation and treatment in a hospital setting. There are 7 items for anxiety and 7 items for depression. A 4 point scale (0-3) is used for each. "0" indicates a negative response and "3" the highest positive response. The total score is the sum of the anxiety and depression scores. 0-7= non case, 8-10= borderline case, 11+= case.
Difference in Spinal cord independence measurement scale (SCIM) between groups | At admission and at discharge from hospital or 24 weeks, whichever is earlier.
  This scale assesses the independence of a spinal cord injury patient in key areas of self-care, respiration and mobility. There are 4 items in 'Self-care', 4 items in 'Respiration and Sphincter management', and 9 items in 'Mobility'. Score of each section is obtained by adding the individual item scores. Total score is 100 obtained from adding the scores of the 3 sections.
Difference in Walking Index for Spinal Cord Injury II (WISCI II) between groups | At admission and at discharge from hospital or 24 weeks, whichever is earlier.
  The Walking Index for Spinal Cord Injury. It corporates the extent and nature of assistance requires for walking in spinal cord injury patients. It is an ordinal scale consisting of 21 levels from "0" being unable to walk with all possible support to "20" being "able to walk with no assistive device, brace or support". The score corresponding to the person's ambulatory status is taken.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Heath and Neurosciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No